CLINICAL TRIAL: NCT03892226
Title: Cardiomyocyte Injury Following Acute Ischemic Stroke
Acronym: CORONA-IS
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. med. Jan Friedrich Scheitz, Principal Investigator, Clinician Scientist, Charite University, Berlin, Germany
Other Study IDs: EA4/123/18
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Ischemic; Cardiac Complication
Keywords: stroke; stroke-heart syndrome; troponin; myocardial stunning; acute coronary syndrome; periodic repolarization dynamics; cardiac complications
MeSH Terms: conditions — Ischemic Stroke; Stroke; Myocardial Stunning; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1, no myocardial injury: normal troponin level (hs-troponin T ≤ 99. percentile, i.e. 14ng/ml)
- 2, chronic myocardial injury: elevated, but stable troponin level; (hs-troponin T> 99. percentile and rise/fall ≤ 20% in the control)
- 3, acute myocardial injury: dynamic troponin elevation; (hs-troponin T> 99. percentile and rise/fall >20% in the control)

SUMMARY:
The primary goal of the CORONA-IS study is to characterize stroke-associated acute myocardial injury (elevated hs-cardiac troponin) using different diagnostic examinations in order get a better understanding of it's underlying pathomechanisms.

DETAILED DESCRIPTION:
Myocardial injury (i.e. elevated cardiac troponin levels) is a frequent cardiac complication during the first few days after an ischemic stroke and is associated with a poor functional outcome. Myocardial injury represents one essential part of a broad spectrum of cardiac complications ranging to severe arrhythmia or heart failure. There is evidence that, in the majority of patients, the underlying mechanism of stroke-associated myocardial injury is not coronary-mediated myocardial ischemia but rather stroke-induced functional and structural interference in the central autonomic network. The investigators hypothesize that this causes a dysregulation of normal neuronal cardiac control leading to myocardial edema and stunning ('Stroke-Heart-Syndrome') CORONA-IS is a prospective, observational, single-centered cohort study that will recruit 300 patients with acute ischemic stroke. According to serial high sensitivity cTn levels during the first 24h after admission, patients will be assigned to three groups (no myocardial injury, chronic myocardial injury, acute myocardial injury). Study procedures include cardiovascular MRI and transthoracic echocardiography to visualize (transient) cardiac dysfunction and provide detailed tissue characterization, 20-minute Holter-monitoring with an analysis of specific autonomic markers, and a systematic bio-banking to study further mechanisms such as altered microRNA signatures. A follow-up for cardiovascular events will be conducted one year after enrolment to study long-term effects of stoke-associated myocardial injury.

The aim of the CORONA-IS study is to develop a better understanding of the characteristics and the pathophysiology of stroke-induced acute myocardial injury ('Stroke-Heart-Syndrome') in order to identify patients at risk and improve diagnostic and therapeutic procedures.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* diagnosis of acute ischemic stroke and hospital admission within 48h after onset of the symptoms
* diagnosis based on visible DWI-lesion in MRI
* written informed consent by participant
* repeated measurement of high sensitive Troponin T within 24h of admission (hs-troponin T, Roche Elecsys®, 99. percentile, upper reference limit=14ng/l)

Exclusion Criteria:

* Pregnancy and / or breast-feeding.
* Impaired renal function (eGFR < 30 ml/min/1,73 m^2)
* Contraindications to undergo MRI (i.e., mechanic heart valve, cardiac pacemaker, etc.)
* Persistent or permanent atrial fibrillation
* ST- elevation myocardial infarction
* History of coronary artery bypass surgery or percutaneous trans-luminal coronary angioplasty (PTCA) ≤ four weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with acute ischemic stroke admitted to the hospital's stroke unit will be systematically screened for eligibility
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of myocardial edema without late gadolinium enhancement (native T1, T2 mapping) | within five days of admission to hospital
  diagnosed in cardiovascular MRI (CMR), conducted at the fourth/fifth day after onset of the ischemic stroke
Rate of myocardial fibrosis with late Gadolinium enhancement (LGE) and acute edema in CMR | within five days of admission to hospital
  Rate of myocardial fibrosis with LGE and acute edema in CMR, suggesting a recent myocardial infarction (<1 month). CMR conducted at the fourth/fifth day after onset of the ischemic stroke.
Rate of signs of left ventricular dysfunction in the CMR | within five days of admission to hospital
  Rate of signs of left ventricular dysfunction in the cardiac MRI (i.e. reduced ejection fraction, end diastolic left ventricular volume, longitudinal strain rate). CMR conducted at the fourth/fifth day after onset of the ischemic stroke.
Rate of acute disturbance of microcirculation | within five days of admission to hospital
  Rate of acute disturbance of microcirculation (measurement on the basis of oxygen extraction in cardiac MRI). CMR conducted at the fourth/fifth day after onset of the ischemic stroke.
Rate of impaired left ventricular function and transient impaired left ventricular function in transthoracic echocardiography | within seven days of admission to hospital
  Rate of impaired left ventricular function (ejection fraction <50%, reduced global longitudinal strain etc.) in the transthoracic echocardiography as well as higher rate of transient left ventricular dysfunction detected in repeated transthoracic echocardiography (TTE). The TTE will be conducted at the first day after enrolment as well as at the day before discharge or five days after the first TTE respectively.

SECONDARY OUTCOMES:
Rate of pathologic Periodic Repolarization Dynamics (PRDs) and Deceleration Capacity (DC) | within seven days of admission to hospital
  Rate of Periodic Repolarization Dynamics (PRDs) and Deceleration Capacity (DC) in the 20 minutes Holter ECG as sign of enhanced sympathetic activity (PRD> 5.75 deg^2, DC ≤2.5 ms).
Difference in specific microRNA pattern in participants with myocardial damage induced by acute ischemic stroke | within seven days of admission to hospital
  Analysis of circulating microRNA pattern via next generation Sequencing in patient's blood samples.
Mortality | at one week and twelve months after the initial event
  mortality (rate of deaths) will be recorded during the stay in hospital as well as after twelve months
Functional outcome | at baseline, at seven days after baseline (or at day of discharge from hospital if <7d, respectively) and at twelve months after the initial event
  functional outcome will be evaluated using the 'modified Rankin scale' (range from 0 = no symptoms to 6 = death; favorable outcome defined as 0 or 1 in the modified Rankin scale)
Rate of cardiovascular events | at one week and at twelve months after the initial event
  cardiovascular events include new stroke, transient ischemic attack and myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Jan Scheitz, PD Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheitz JF, Nolte CH, Doehner W, Hachinski V, Endres M. Stroke-heart syndrome: clinical presentation and underlying mechanisms. Lancet Neurol. 2018 Dec;17(12):1109-1120. doi: 10.1016/S1474-4422(18)30336-3. Epub 2018 Oct 26. PMID 30509695
- [Background] Mochmann HC, Scheitz JF, Petzold GC, Haeusler KG, Audebert HJ, Laufs U, Schneider C, Landmesser U, Werner N, Endres M, Witzenbichler B, Nolte CH; TRELAS Study Group. Coronary Angiographic Findings in Acute Ischemic Stroke Patients With Elevated Cardiac Troponin: The Troponin Elevation in Acute Ischemic Stroke (TRELAS) Study. Circulation. 2016 Mar 29;133(13):1264-71. doi: 10.1161/CIRCULATIONAHA.115.018547. Epub 2016 Mar 1. PMID 26933082
- [Background] Rizas KD, Hamm W, Kaab S, Schmidt G, Bauer A. Periodic Repolarisation Dynamics: A Natural Probe of the Ventricular Response to Sympathetic Activation. Arrhythm Electrophysiol Rev. 2016 May;5(1):31-6. doi: 10.15420/aer.2015:30:2. PMID 27403291
- [Background] Stengl H, Ganeshan R, Hellwig S, Blaszczyk E, Fiebach JB, Nolte CH, Bauer A, Schulz-Menger J, Endres M, Scheitz JF. Cardiomyocyte Injury Following Acute Ischemic Stroke: Protocol for a Prospective Observational Cohort Study. JMIR Res Protoc. 2021 Feb 5;10(2):e24186. doi: 10.2196/24186. PMID 33544087
- [Background] Scheitz JF, Stengl H, Nolte CH, Landmesser U, Endres M. Neurological update: use of cardiac troponin in patients with stroke. J Neurol. 2021 Jun;268(6):2284-2292. doi: 10.1007/s00415-020-10349-w. Epub 2020 Dec 29. PMID 33372247
- [Derived] Rosso M, Stengl H, Ganeshan R, Hellwig S, Klammer MG, von Rennenberg R, Bohme S, Nolte CH, Audebert HJ, Endres M, Kasner SE, Scheitz JF. Sex Differences in Outcomes of Acute Myocardial Injury After Stroke. J Am Heart Assoc. 2024 Mar 5;13(5):e032755. doi: 10.1161/JAHA.123.032755. Epub 2024 Feb 27. PMID 38410952